CLINICAL TRIAL: NCT04039581
Title: Short-Term Effects of Kinesio Taping® on Pain and Functionality in Patients with Cervical Spine Surgery
Brief Title: KT® in Patients with Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Marmara University
Record Dates: First submitted 2019-07-24; First posted 2019-07-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pain; Cervical Spinal Stenosis; Disc, Herniated; Cervical Spondylosis
Keywords: Kinesio Tape; Pain; Functionality; Cervical Spine Surgery
MeSH Terms: conditions — Pain; Intervertebral Disc Displacement; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Kinesio Taping and Conventional treatment (Experimental): The number of participants in this group is anticipated to be 30. The treatment method for this group is the conventional treatment + KT (Kinesio Taping) (Space Correction).
  In the conventional treatment therapeutic exercises (active and passive Range Of Motion (ROM) and strengthening exercise of the neck and shoulder) and TENS (Transcutaneous electrical nerve stimulation) applications on the painful area, every day and 2 channels with 4 electrodes in the acute period (first 72 hours) will be applied. These exercises will be taught to participants from the first treatment session and will be performed under the supervision of a physiotherapist. In KT technique, while participants are sitting on the edge of the bed, the shoulder area will be depressed and I banding will be done by applying 25-50% tension horizontally in this position on the upper trapezius muscle.
  Interventions: Other: Kinesio Taping; Other: Conventional treatment
- Group 2: Conventional treatment (Active Comparator): The number of participants in this group are anticipated to be 30. This group will be receiving only conventional treatment. In the conventional treatment therapeutic exercises (active and passive range of motion (ROM) and strengthening exercise of the neck and shoulder) and TENS (Transcutaneous electrical nerve stimulation) applications on the painful area, every day and 2 channels with 4 electrodes in the acute period (first 72 hours) will be applied. These exercises will be taught to participants from the first treatment session and will be performed under the supervision of a physiotherapist.
  Interventions: Other: Conventional treatment
- Group 3: Kinesio Taping (Active Comparator): The number of participants in this group are anticipated to be 30. This group will be receiving only Kinesio Taping (Space Correction). In kinesio taping technique while participants are sitting on the edge of the bed, the shoulder area will be depressed and I banding will be done by applying 25-50% tension horizontally in this position on the upper trapezius muscle.
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio Taping (Space Correction).
  Arms: Group 1: Kinesio Taping and Conventional treatment; Group 3: Kinesio Taping
Other: Conventional treatment — Therapeutic exercises (active and passive range of motion (ROM) and strengthening exercise ) and TENS (Transcutaneous electrical nerve stimulation) applications
  Arms: Group 1: Kinesio Taping and Conventional treatment; Group 2: Conventional treatment

SUMMARY:
Aim of the study was to investigate the effect of Kinesio taping application on upper trapezius muscle after cervical spine surgery.

DETAILED DESCRIPTION:
Patients will be randomly divided into three groups. The first group will receive conservative treatment and Kinesio Taping application. The second group will receive conservative treatment and the third group will receive only Kinesio taping application. The treatment procedure will continue for post-operatively three days and assessments will be done four times; before the surgery, post-operative 1st day, postoperative 3rd day and two weeks after surgery. Data will be recorded on patient assessment file and transferred to the computer. Data analysis will be performed with SPSS.22.

ELIGIBILITY:
Inclusion Criteria:

* To be voluntary participation in the study,
* Aged 25-75 years old,
* To be diagnosed with cervical disc herniation, cervical stenosis and cervical spondylolisthesis
* No mental problem, sensory or motor aphasia in order to understand and answer the evaluation questions correctly.

Exclusion Criteria:

* History of surgery,
* Allergic reaction to kinesio taping,
* Primary or metastatic neoplasm in cervical spine,
* History of different treatment for neck pain during the study period,
* Individuals with any congenital deformity in the spine,
* Having any rheumatologic, neurological and orthopedic disease.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change from baseline to two weeks after the surgery
  Neck pain intensity will be assessed with Visual Analog Scale (VAS).The VAS is usually a horizontal line, 10 cm in length, anchored by word descriptors at each end with "No Pain" (score of zero) on the left side up to "pain as bad as it could be" or the "worst imaginable pain" (Score of 100 [100-mm scale]) on the right side.The patient was asked to mark the line point that represented his or her current pain.
Pain pressure threshold | Change from baseline to two weeks after the surgery
  Pain pressure threshold of the trapezius muscle will be evaluated by digital pressure algometry. In the process, three measurements will be taken and the average value will be taken as reference.

SECONDARY OUTCOMES:
Range of Motion (ROM) | Change from baseline to two weeks after the surgery
  Range of motion will be measured with a goniometer. The goniometer is valid and reliable tool.
Disability | Change from baseline to two weeks after the surgery
  Disability will be assessed with Neck Pain and Disability Scale (NPAD). Turkish version of the Neck Pain and Disability Scale is including 20 items which measure the intensity of neck pain and related disability. Item scores range from 0 to 5. Each item has a 10-cm visual analog scale. It has six major divisions divided into equal intervals by vertical bars. The questions are investigating the relationship between neck pain severity and pain on occupational life, recreational activities, social and functional aspects of living, and emotional factors. High scores indicate serious disabilities.
Health Related Quality of Life Score | Change from baseline to two weeks after the surgery
  Quality of life will be assessed with Short Form-36 (SF-36).The SF-36, It generates 8 subscales and two summary scores.The 8 subscales are; physical functioning, role limitations due to physical health, role, limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, bodily pain, general health perceptions. The two summary scores are the physical component summary and the mental component summary. Scoring the SF-36 consists of 36 items. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Functionality Score | Change from baseline to two weeks after the surgery
  The functionality will be assessed with Upper Extremity Functional Index-15 (UEFI-15). The UEFI-15 consists of 15 questions on a 5- point rating scale assessing level of difficulty in performing activities of daily living using the upper extremities. 0 indicates extreme difficulty while 4 indicates no difficulty wit a task. The scores given to the 15 questions are added to give the highest possible score of 60 and the lowest possible score is 0. A lower score indicates that the person is reporting increased difficulty with the activities as a result of their upper limb functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba KURU ÇOLAK, Study Director — Marmara University
Locations (1):
- Bahçeşehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartleson JD. Low Back Pain. Curr Treat Options Neurol. 2001 Mar;3(2):159-168. doi: 10.1007/s11940-001-0051-4. PMID 11180753
- [Background] Gonzalez-Iglesias J, Fernandez-de-Las-Penas C, Cleland JA, Huijbregts P, Del Rosario Gutierrez-Vega M. Short-term effects of cervical kinesio taping on pain and cervical range of motion in patients with acute whiplash injury: a randomized clinical trial. J Orthop Sports Phys Ther. 2009 Jul;39(7):515-21. doi: 10.2519/jospt.2009.3072. PMID 19574662
- See also: Low Back Pain — https://www.ncbi.nlm.nih.gov/pubmed/11180753
- See also: hort-term effects of cervical kinesio taping on pain and cervical range of motion in patients with acute whiplash injury: a randomized clinical trial. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Short-term+effects+of+cervical+kinesio+taping+on+pain+and+cervical+range+of+motion+in+patients+with+acute+whiplash+injury%3A+a+randomized+clinical+trial.